CLINICAL TRIAL: NCT05724394
Title: A Feasibility Randomized Controlled Trial of Culturally Adapted Getting Better Bite-by-Bite (Ca-GBBB)Intervention for Individuals With Eating Disorders in Pakistan
Brief Title: Feasibility Trial of Getting Better Bite by Bite for Eating Disorders
Acronym: CaGBBB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PILL-GBBB-ED
Record Dates: First submitted 2022-12-09; First posted 2023-02-13 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Eating Disorders; Bulimia Nervosa; Binge-Eating Disorder
Keywords: Getting better bite by bite (GBBB); Culturally Adapted Intervention; Low resource settings; Pakistan; Eating Disorders; Feasibility Study
MeSH Terms: conditions — Feeding and Eating Disorders; Bulimia Nervosa; Binge-Eating Disorder | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Feasibility Randomized Controlled Trial with participants randomized into two trial arms
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ca-GBBB arm (Experimental): The Ca-GBBB strongly focuses on enhancing participant's motivation and belief in their ability to change. The intervention will be comprised of 16-week training program delivered over four months. Sessions will be delivered weekly and each session will last about 45-50 minutes. All sessions will be delivered by master level psychologist. The manual will be translated to Urdu giving special consideration to cultural adaptation of phrases and concepts to reflect Pakistani culture. Additionally, culturally appropriate case scenarios will be incorporated and a consensual view to addressing cultural factors such as gender role, financial difficulties will be taken into consideration. The time and venue of session will be decided prior according to participant convenience.
  Interventions: Other: Culturally Adapted Getting Better Bite By Bite (Ca-GBBB) intervention
- Treatment As Usual (No Intervention): Treatment as Usual (TAU) group will receive routine care and their follow up will be done at 4-month post-randomization.

INTERVENTIONS:
Other: Culturally Adapted Getting Better Bite By Bite (Ca-GBBB) intervention — The Ca-GBBB strongly focuses on enhancing participant's motivation and belief in their ability to change. The intervention will be comprised of 16-week training program delivered over four months.
  Arms: Ca-GBBB arm

SUMMARY:
This is a mixed method feasibility randomized controlled trial to explore the feasibility and acceptability of therapist delivered, culturally adapted, manualized Ca-GBBB intervention for Eating Disorders (EDs) - Bulimia Nervosa (BN) and Bing Eating Disorder (BED) in Pakistan.

DETAILED DESCRIPTION:
Evidence on psychological management of eating disorders in low and middle income countries ( LMICs) is limited, and non-existent in Pakistan. A Cognitive Behaviour Therapy (CBT) based guided self-help manual "Getting Better Bite by Bite: A Survival Kit for Sufferers of Bulimia Nervosa and Binge Eating Disorders" (GBBB), has found to be feasible and acceptable for patients with BN.

Quantitative phase of this research aims to determine if the culturally adapted GBBB (Ca-GBBB) programme is feasible and acceptable for individuals with Eating disorders- BN and BED compared to treatment as usual.

The qualitative part of the study will include focus groups and in-depth digitally recorded one-to-one interviews with participants by trained qualitative researchers at two time points both before and after the intervention. These focus groups and in-depth interviews will continue till the data saturation is achieved. Moreover, in-depth digitally-recorded interviews with stakeholders (nutritionists, dietitian, educationist, therapists, health professionals, etc) will also be conducted by trained researchers.

ELIGIBILITY:
Inclusion Criteria:

1. Age18 years
2. Screen positive on the Binge Eating Screening Questionnaire and/or Bulimic Investigatory test, Edinburgh
3. Residents of the study catchment area
4. Able to provide informed consent

Exclusion Criteria:

1. Aged under 18
2. Presence of any severe mental or physical illness that would prevent individual from participating in the intervention and or assessments.
3. Temporary resident unlikely to be available for follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-04-28 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment and attrition Logs | One year's time
  The parameters feasibility of undertaking the trial of intervention will include the recruitment rate (the number of patients referred/approached, proportion of those who consented out of all the eligible patients with BED and/or BN disorder referred from and approached at the recruitment sites) (The success criterion of feasibility will be to recruit > 50% of eligible participants) and the attrition rate (the number of patients withdrawn out of those who consented to participate).
Intervention Log | During 4-month intervention period.
  Feasibility of the intervention delivery: Duration of each session and completed feedback forms. This will be assessed by keeping record of whether the Ca-GBBB is delivered, received and enacted as intended.
Attendance logs | From baseline to 4-month follow up
  Therapy logs will include each participant's attendance in a session. This will give information about acceptability of intervention. mean attendance rate of >70% i.e. at least 11 sessions, will indicate that the intervention is acceptable for the participants
Client Satisfaction Questionnaire | From baseline to 4-month follow up
  Tolerability of the intervention is defined as the ability to endure the intervention. Items on Client Satisfaction Questionnaire are scored on a four-point Likert scale from 1 (low satisfaction) to 4 (high satisfaction), with different descriptors for each response point. Totals range from 8 to 32; with higher scores indicating greater satisfaction.

SECONDARY OUTCOMES:
The Bulimic Investigatory Test, Edinburgh | Change in score from baseline to 4-month follow-up.
  The BITE is a 33-item self-rating scale (Henderson and Freeman 1987). It consists of two subscales: The Symptom Scale (30 items), which measures the degree of symptoms and the Severity Scale (3 items), which provides an index of the severity as defined by the frequency of binge-eating and purging behavior. The total score for all the questions gives a "symptom score" - a score of 15 or above indicate that the individuals has a lot of thoughts and attitudes consistent with eating disorders. The toral score of question 6, 7 and 27 will give a severity index - a score of 5 or above signifies an eating disorder
Binge-Eating Disorder Screener | Change in score from baseline to 4-month follow-up
  The 7-item Binge-Eating Disorder Screener (BEDS-7), a brief screener for BED, can assist physicians in identifying patients who may have BED. Those with a score of 2-3 are considered mildly at risk of BED, a score of 4-5 is determined to be moderately at risk for BED, and a score of 6 indicates severely at risk for BED
The Sick, Control, One, Fat, Food | Change in score from baseline to 4-month follow-up
  5 item questionnaire that covers the main three domains which are anorexia nervosa, bulimia nervosa, or other eating disorders. Each yes answer means 1 point and if the interviewee gets 2 points it reveals that he/she has anorexia nervosa or bulimia.
Eating Disorder Examination Questionnaire | Change in score from baseline to 4-month follow-up
  a 28-item self-reported questionnaire adapted from the semi-structured interview Eating Disorder Examination (EDE) and designed to assess the range and severity of features associated with a diagnosis of eating disorder using 4 subscales (Restraint, Eating Concern, Shape Concern and Weight Concern) and a global score. Higher scores on the global scale and subscales denote more problematic eating behaviours and attitudes. A cut-off of 4 on the global score is generally used as clinically significant
Kessler Psychological Distress Scale | Change in score from baseline to 4-month follow-up
  It is used to measure psychological distress. It's a 10 item scale measuring emotional states with a 5 level response scale. Scores will range from 10 to 50. Low scores indicate low levels of psychological distress and high scores indicate high levels of psychological distress. score 10 - 19 Likely to be well, 20 - 24 Likely to have a mild disorder, 25 - 29 Likely to have a moderate disorder and 30 - 50 Likely to have a severe disorder
Beck Scale for Suicidal Ideation | Change in score from baseline to 4-month follow-up
  The BSS is a 21-item measure that will be used to assess the frequency and intensity of suicidal thoughts. Each item is scored based on an ordinal scale from 0 to 2 and the total score is 0 to 38. Individuals answer to the first 5 items which is excerpted. If individual's answer to the fifth item is positive (scores 1 and 2), he/she answers the rest of the items and otherwise the questionnaire is completed. No cut- point is used to categorize the scores
Beck Depression Inventory | Change in score from baseline to 4-month follow-up
  The BDI is a 29 item questionnaire that will be used to measure severity of depression. Score 1-10 are considered normal, 11-16 Mild mood disturbance, 17-20 Borderline clinical depression, 21-30 Moderate depression, 31-40 Severe depression over 40 Extreme depression
Oslo- 3 Social Support Scale | Change in score from baseline to 4-month follow-up
  O3SSS will be used to assess the relationship with friends, family and neighbors. The sum score ranges from 3 to 14, with high values representing strong levels and low values representing poor levels of social support. The OSSS-3 sum score can be operationalized into three broad categories of social support: a) 3-8 poor social support, b) 9-11 moderate social support, c) 12-14 strong social support
Client Satisfaction Questionnaire | Change in score from baseline to 4-month follow-up
  Participant satisfaction with services will be assessed using the Client Satisfaction Questionnaire (CSQ). Scores are summed across items once. Items 2, 4, 5, and 8 are reverse scored. Total scores range from 8 to 32, with the higher number indicating greater satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Lahore site, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The anonymised data will be shared on request
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Result] Atwood ME, Friedman A. A systematic review of enhanced cognitive behavioral therapy (CBT-E) for eating disorders. Int J Eat Disord. 2020 Mar;53(3):311-330. doi: 10.1002/eat.23206. Epub 2019 Dec 16. PMID 31840285
- [Derived] Khaliq A, Muazzam A, Rafique R, Kiran T, Ahmed A, Suleheria I, Chaudhry N, Husain N. A feasibility randomized controlled trial of culturally adapted Getting Better Bite-by-Bite (Ca-GBBB) intervention for individuals with eating disorders in Pakistan. J Eat Disord. 2024 Jul 17;12(1):100. doi: 10.1186/s40337-024-01038-4. PMID 39020405